CLINICAL TRIAL: NCT06809257
Title: Effect of Exercise on MiR-126 in Individuals With Prediabetes: A Randomized Controlled Trial
Brief Title: Effect of Exercise on MiR-126 in Individuals With Prediabetes
Acronym: EMiR-126-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Elif Yıldırım Ayaz, Assoc. Prof. Dr., Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EMiR-126-PD; Saglik Bilimleri University (Other: Saglik Bilimleri University)
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Prediabetes; microRNA; Exercise
Keywords: MiR-126; Exercise; Prediabetes; MicroRNA
MeSH Terms: conditions — Prediabetic State; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator): Individuals in the intervention group were included in a planned aerobic exercise program for 12 weeks.This program was carried out under the supervision of specialist doctors, with the help of sports trainers and physiotherapists, and participants were given 60 minutes of moderate-intensity (50-70% of their maximum heart rate) aerobic exercise three days a week.
  Interventions: Behavioral: Exercise
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Exercise — 12 week moderately aerobik exercise
  Arms: Exercise

SUMMARY:
This study aims to investigate the effect of a structured exercise program on microRNA-126 (miR-126) expression in individuals with prediabetes.

DETAILED DESCRIPTION:
This study aims to investigate the effect of a structured exercise program on microRNA-126 (miR-126) expression in individuals with prediabetes. The hypothesis of our study is that regular aerobic exercise will increase miR-126 expression. Determining the effect of exercise on miR-126 in individuals with prediabetes will contribute to the elucidation of the pathways through which exercise is effective in prediabetes via epigenetic mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were newly diagnosed with prediabetes according to the Oral Glucose Tolerance Test (OGTT) and/or HbA1C criteria
* between the ages of 18-60
* were physically inactive (Level 1 according to the International Physical Activity Questionnaire)
* were motivated to exercise
* Individuals who had no obstacle to exercise as a result of the evaluation made by a cardiologist (ECG, exercise ECG test, etc.)
* and who did not show a change in body weight of more than ±2.5 kg in the last six months were included in the study.

Exclusion Criteria:

* presence of serious medical conditions (e.g. advanced cancer, major neurological or endocrine disorders, respiratory failure)
* current cardiovascular disease, BMI <19 kg/m²
* history of metformin use within the last 6 months
* receiving hormone replacement therapy
* life expectancy less than one year
* HIV positivity
* substance use
* or orthopedic and cognitive disorders that may prevent exercise

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Delta CT mir-126 | 1 week
  Ct (cycle threshold) values for miR-126 and miR-16-5p were used for analysis. ΔCt and ΔΔCt values were calculated as follows, and expression levels were analyzed using the 2-ΔΔCt method:
  ∆Ct = Ct (gene of interest) - Ct (housekeeping gene) ΔΔCt = ∆Ct (treated sample) - ∆Ct (untreated sample) Higher ΔCt values indicate lower expression levels.

SECONDARY OUTCOMES:
BMI | 1 day
  The BMI is calculated by dividing an adult's weight in kilograms by their height in metres squared.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, Principal Investigator — Sultan 2. Abdülhamid Han Training and Research Hospital
Locations (1):
- Sultan 2. Abdülhamid Han Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No